CLINICAL TRIAL: NCT06067776
Title: A Phase I Study of Osimertinib, Cetuximab, and Tucatinib in Advanced EGFR-Mutant NSCLC With Acquired Resistance to Osimertinib
Brief Title: Osimertinib, Cetuximab, and Tucatinib for the Treatment of EGFR-Mutant Stage IV or Recurrent Non-small Lung Cell Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonathan Riess (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jonathan Riess, Sponsor-Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#298; NCI-2022-04431 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#298 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cetuximab; osimertinib; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tucatinib, osimertinib, cetuximab) (Experimental): Patients receive tucatinib 200mg orally BID, osimertinib 80mg orally daily, and cetuximab 250mg/m^2 IV every 2 weeks of a 28-day cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Osimertinib; Drug: Tucatinib

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: ERBITUX
Drug: Osimertinib — Given PO
  Other Names: TAGRISSO
Drug: Tucatinib — Given PO
  Other Names: TUKYSA

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of osimertinib, cetuximab, and tucatinib in treating patients with EFGR-mutant non-small cell lung cancer that is stage IV or has come back (recurrent). Osimertinib and tucatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

Cetuximab is a chimeric human/mouse IgG1 monoclonal antibody that targets epidermal growth factor receptor (EGFR), a receptor overexpressed in many types of cancer, and may interfere with the ability of tumor cells to grow and spread. Giving osimertinib, cetuximab, and tucatinib may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE :

I. To estimate the maximum tolerated dose (MTD) of osimertinib, cetuximab, and tucatinib in participants with EGFR-mutant non-small cell lung cancer (NSCLC) who have acquired resistance to EGFR-tyrosine kinase inhibitor (TKI).

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of osimertinib, cetuximab, and tucatinib in participants with EGFR-mutant NSCLC who have acquired resistance to EGFR-TKI.

II. To obtain preliminary assessment of anti-tumor activity of osimertinib, cetuximab, and tucatinib in participants with EGFR-mutant NSCLC who have acquired resistance to EGFR-TKI (osimertinib).

III. To obtain preliminary assessment of anti-tumor activity of osimertinib, cetuximab, and tucatinib in the dose expansion cohort of participants with EGFR-mutant NSCLC who progressed on first-line osimertinib and do not have non-ERBB bypass tract mechanisms of resistance, including a subset of participants positive for HER2 aberrant signaling as determined by immunohistochemistry (IHC), fluorescence in situ hybridization (FISH) and/or next generation sequencing (NGS).

OUTLINE:

This is a dose-escalation study of tucatinib and cetuximab. Patients receive tucatinib 200mg orally BID, osimertinib 80mg orally daily, and cetuximab 250mg/m^2 IV every 2 weeks of a 28-day cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at 30 days and every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Stage IV or recurrent/metastatic histologically confirmed non-small cell lung cancer (NSCLC).
* NSCLC must harbor at least one of the following EGFR activating mutations: Exon 21 L858R, Exon 19 deletion, Exon 18 G719X, Exon 21 L861Q, Exon 20 S768I.
* For patients in the dose escalation cohort, patients must have progressed on any prior EGFR-Tyrosine Kinase Inhibitor (TKI) and if T790M positive must have also progressed on osimertinib. Participants in the dose expansion cohort must have had progressive disease as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) version (v)1.1 criteria on osimertinib as first-line therapy.
* 4. Participants in the dose expansion cohort must be negative for clinically significant non-ERBB bypass tract resistance such as MET amplification, BRAF mutation, RAS-RAF-MAPK alteration, ALK fusion, RET fusion by a Clinical Laboratory Improvement Amendments (CLIA) (performed after progression on prior EGFR-TKI; if any questions please consult with the Principal Investigator). A defined subset of patients in the expansion cohort will have human epidermal growth factor receptor (HER2) aberrant signaling as putative resistance to osimertinib with overexpression/amplification (or more rarely HER2 Exon 20 insertion mutation) as determined by IHC (3+ IHC) or FISH (HER2/CEP17 > 2.2 or HER2 copy number > 6) or NGS for HER2 mutation.
* Adequate archival tissue from a biopsy performed after progression of disease on previous osimertinib (or last EGFR-TKI for dose escalation cohort) or willingness to consent for a fresh tumor biopsy.
* Participants must have measurable disease by RECIST 1.1, by positron emission tomography/computed tomography (PET/CT) or CT imaging within 28 days prior to registration. The CT from a combined PET/CT may be used only if it is of diagnostic quality.
* Men and women >=18 years of age at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy greater than 3 months.
* Absolute neutrophil count >= 1.5 x 10^9/L.
* Platelets >= 100 x 10^9/L.
* Hemoglobin >= 9 g/dL.
* Serum albumin >= 2.5 g/dL.
* Bilirubin =< 1.5 x the upper limit of normal (ULN).
* Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate transaminase (AST) =< 2.5 x ULN.
* Potassium within institutional normal limits.
* Magnesium within institutional normal limits.
* Coagulation parameters of international normalized ratio (INR) < 1.5 and partial thromboplastin time (PTT) < 30 seconds.
* Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 50 mL/min (per the Cockcroft-Gault formula).
* If brain metastases are present, they must be stable and asymptomatic. Participants on corticosteroids for brain metastases are excluded.
* Left ventricular ejection fraction 50% or more on echocardiogram or multigated acquisition scan.
* Individuals of child-bearing potential must test negative for pregnancy =< 14 days prior to receiving first dose of study medication based on a serum pregnancy test and agree to use 2 methods of birth control or abstain from heterosexual activity during the study and for 6 months following the last dose of the study drug(s), whichever is longer; or be of non- childbearing potential. Non-childbearing potential is defined as (by other than medical reasons) * >= 45 years of age and has not had menses for greater than 2 years. * Amenorrheic for < 2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation. *Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed (of the actual procedure or confirmed by an ultrasound). Tubal ligation must be confirmed (of the actual procedure) otherwise the participant must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 6 months after the last dose of study therapy.
* Ability to swallow pills.
* Ability to understand and willingness to sign an informed consent form.
* Ability to adhere to the study visit schedule and protocol requirements.
* Participants previously on osimertinib allowed to continue prior to initiating study.

Exclusion Criteria:

* History of pneumonitis requiring steroids, including history of radiation-induced pneumonitis.
* Known or suspected leptomeningeal disease as documented by the investigator. Stable asymptomatic brain metastases not requiring steroids is allowed; radiation for brain metastases is allowed as long as there is a two-week washout period prior to starting study treatment.
* Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding central nervous system (CNS)-directed therapy.
* The participant has a known allergy / history of hypersensitivity reaction to any of the treatment components (including any ingredient or similar ingredient used in the product formulations) or red meat.
* History of tick bite or any other contraindication to one of the administered treatments.
* History of arterial or venous thromboembolism within 3 months prior to study enrollment. Participants with a history of venous thromboembolism beyond 3 months prior to study enrollment can be enrolled if they are appropriately treated with low molecular weight heparin or direct oral anti-coagulants.
* History or evidence of current clinically relevant coronary artery disease >= Grade III by the Canadian Cardiovascular Society Angina Grading Scale or uncontrolled congestive heart failure of current > Class III as defined by the New York Heart Association.
* The participant has experienced myocardial infarction within 6 months prior to study enrollment.
* The participant has a history of clinically significant ventricular arrhythmia, cardiac arrest, or torsades de pointes.
* The participant has high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
* The participant has uncontrolled or poorly controlled hypertension (>180 mmHg systolic or > 130 mmHg diastolic.
* Use of a strong cytochrome P450 CYP2C8 inhibitor within 5 half-lives of the inhibitor or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to the first dose of study treatment.
* The participant is pregnant or breast feeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.
* The participant has any ongoing or active clinically significant infection, including known active tuberculosis or known ongoing or active infection with the human immunodeficiency virus.
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination.
* Any condition that would prohibit the understanding or rendering of informed consent.
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial.
* Radiation within 14 days before beginning study drugs.
* Prior EGFR monoclonal antibody treatment (i.e., necitumumab or cetuximab) or HER2 directed treatment (i.e., trastuzumab deruxtecan) for dose expansion only.
* Any systemic therapy within 3 weeks of enrollment with the exception of EGFR-TKI. * Platinum-based chemotherapy or other lines of intervening systemic therapy after progression on osimertinib or EGFR TKIs is allowed but must be completed no later than 3 weeks before study enrollment.
* Prior EGFR-TKI (if not osimertinib) must be discontinued at least 7 days prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | First dose through cycle 1 (each cycle is 28 days)
  The occurrence of a dose-limiting toxicity in participants receiving the combination of osimertinib, cetuximab, and tucatinib.

SECONDARY OUTCOMES:
Incidence of adverse events | First dose through 30 days post last dose
  Number of participants experiencing adverse events (AEs), both non treatment related and treatment related, classified by severity and graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.
Objective response rate (ORR) | First dose through progression or end of study treatment, whichever occurs first, assessed up to 10 months
  Objective response rate (ORR), assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Progression-free survival (PFS) | Up to 2 years post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Riess, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States